CLINICAL TRIAL: NCT06645912
Title: Effect of High Protein Nutritional Supplementation on Nutritional Status, Functional Capacity and Quality of Life in Older Patients With Gastric Cancer Receiving Neoadjuvant Chemotherapy
Brief Title: Effect of High Protein ONS on Older Gastric Cancer Patients Receiving Neoadjuvant Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Binali Yildirim University Mengucek Gazi Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Baran Akagündüz, MD, Associate Proffesor, Erzincan Binali Yildirim University Mengucek Gazi Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-7/14
Record Dates: First submitted 2024-10-12; First posted 2024-10-17 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Locally Advanced Gastric Adenocarcinoma
Keywords: Gastric cancer; Older patients; Oral nutritional supplement
MeSH Terms: conditions — Stomach Neoplasms | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Randomized ıntervantıonal study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONS and standard nutrition support (Experimental): Patients receiving high protein containing oral nutritional supplement with standart nutritional support
  Interventions: Dietary Supplement: oral nutritional supplement
- standart nutrition support (No Intervention): Patients receiving only standart nutritional support

INTERVENTIONS:
Dietary Supplement: oral nutritional supplement — The ONS group received a high-protein ONS providing 18.8 g of protein, 7 g of fat, 28 g of carbohydrates, and 250 calories of energy per 200 mL and medical nutrition therapy. The product is gluten-free and contains lactose, minerals, trace elements, and vitamins . The Control group received only standard nutrition therapy without ONS supplementation.
  Arms: ONS and standard nutrition support

SUMMARY:
This interventional prospective randomized controlled study was conducted to compare the effects of high-protein oral nutritional supplement (ONS) and medical nutritional therapy to medical nutrition therapy alone on nutritional status, quality of life, and physical function capacity after neoadjuvant chemotherapy in patients aged 65 and over with newly diagnosed locally advanced gastric cancer.

DETAILED DESCRIPTION:
This study is a prospective, randomized controlled trial conducted from February 2023 to February 2024, focusing on the effects of high-protein oral nutritional supplementation (ONS) in older patients (aged 65 and over) with newly diagnosed locally advanced gastric cancer undergoing neoadjuvant chemotherapy (NAC).

Study Design:

The trial involved two groups:

Intervention group (ONS group) - Received ONS in addition to standard medical nutrition therapy.

Control group (non-ONS group) - Received only standard medical nutrition therapy without ONS supplementation.

Participants were randomized using computer-aided randomization, with 28 patients in each group. After excluding patients based on specific criteria (e.g., discontinuation of chemotherapy, refusal to consume ONS, or non-compliance with nutrition therapy), 23 patients remained in each group, totaling 46 patients for final analysis.

Patients in the ONS group received a high-protein supplement containing 18.8 g of protein, 7 g of fat, 28 g of carbohydrates, and 250 calories per 200 mL. Both groups received personalized medical nutrition therapy based on their nutritional needs, calculated as 30 kcal/kg/day of energy and 1.5 g/kg/day of protein.

Data Collection and Monitoring:

Data was collected at three key time points:

Baseline (Week 0): Assessments included anthropometric measurements, handgrip strength, food intake records, nutritional status evaluation (Mini Nutritional Assessment), biochemical markers, quality of life (EORTC QLQ-C30), functional status (ADL and IADL), and comorbidity index (Charlson Comorbidity Index).

Mid-Intervention (Week 4): Food intake, MNA, and ONS adherence were re-assessed, with the ONS follow-up form and new anthropometric data collected.

Post-Intervention (Week 8): Final assessments covered all previously mentioned parameters (anthropometry, handgrip strength, MNA, biochemical data, ADL, IADL, EORTC QLQ-C30), alongside an evaluation of compliance and ONS consumption.

Statistical Analysis:

The primary outcome measures were changes in nutritional status, physical function (handgrip strength, ADL, IADL), and quality of life (EORTC QLQ-C30) between baseline and week 8. Secondary outcomes included body composition changes (measured by BIA), adverse events (CTCAE v5.0), and dietary intake analysis using BEBIS software. The intervention's impact was evaluated by comparing pre- and post-intervention changes between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* • Aged 65 years or older.

  * Newly diagnosed histological confirmed locally advanced gastric cancer (Stage IIa to IIIa).
  * Scheduled to receive Neoadjuvant chemotherapy.
  * ECOG performance status of 0-2.
  * Signed informed consent to participate

Exclusion Criteria:

* Severe comorbidities affecting survival within 3 months.

  * Inability to comply with study procedures.
  * Previous gastric surgery or chemotherapy.
  * Metastatic dissease (Stage IV)
  * Poor performance status (ECOG 3-4)
  * Early satge (Stage I)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Change in Mini Nutritional Assessment (MNA) score | Baseline and 8 Weeks
  Unit of Measure: MNA score (Units on a Scale). This will measure changes in nutritional status using the MNA scoring system, which ranges from 0 to 30. A higher score indicates better nutritional status (24-30: normal nutritional status, 17-23.5: at risk of malnutrition, <17: malnourished).
Change in Handgrip Strength | Baseline and 8 Weeks
  Unit of Measure: Kilograms (kg). Measured with a hand dynamometer, the average handgrip strength (kg) will be calculated based on three measurements of the dominant hand.
Change in EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30) score | Baseline and 8 Weeks
  Unit of Measure: QLQ-C30 score (Units on a Scale). The EORTC QLQ-C30 evaluates quality of life across multiple domains, including physical, emotional, and social functioning. Scores range from 0 to 100, with higher scores indicating better quality of life in functioning scales but worse symptoms when higher scores are in symptom scales.
Change in 'Activities of Daily Living' (ADL) Score | Baseline and 8 Weeks
  Unit of Measure: ADL score (Units on a Scale). The ADL scale assesses the patient's ability to perform basic daily tasks, such as bathing, dressing, and feeding. Scores range from 0 to 6, with higher scores indicating better physical function and independence.
Change in 'Instrumental Activities of Daily Living' (IADL) Score | Baseline and 8 Weeks
  Unit of Measure: IADL score (Units on a Scale). The IADL scale evaluates the patient's ability to perform more complex daily tasks, such as managing finances and using transportation. Scores range from 0 to 8, with higher scores reflecting better functional independence.

SECONDARY OUTCOMES:
Change in Body Weight | Baseline and 8 Weeks
  Unit of Measure: Kilograms (kg). Body weight will be recorded in kilograms and tracked over time.
Change in Body Mass Index (BMI) | Baseline and 8 Weeks
  Unit of Measure: kg/m². BMI will be calculated by dividing weight in kilograms by the square of height in meters.
Change in Mid-Upper Arm Circumference | Baseline and 8 Weeks
  Unit of Measure: Centimeters (cm). This anthropometric measurement will be taken with a non-stretchable tape measure.
Change in Calf Circumference | Baseline and 8 Weeks
  Unit of Measure: Centimeters (cm). Calf circumference will also be measured with a tape measure and recorded in centimeters.
Changes in Bioelectrical Impedance Analysis (BIA) | Baseline and 8 Weeks
  Unit of Measure: Percentage (%). BIA will be used to assess body composition, such as body fat percentage and lean mass percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Diğdem DOĞAN AKAGÜNDÜZ, Study Director — Erzincan Mengucek Gazi Research and Training Hospital
Locations (1):
- Erzincan Binali Yıldırım Üniversitesi Mengücek Gazi Eğitim ve Araştırma. Hastanesi, Erzincan, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dogan Akagunduz D, Turker PF, Akagunduz B. Effects of high-protein nutritional supplementation on nutritional status, physical function, and quality of life in older gastric cancer patients receiving neoadjuvant chemotherapy: a randomized trial. Support Care Cancer. 2025 Aug 9;33(9):775. doi: 10.1007/s00520-025-09822-x. PMID 40782206